CLINICAL TRIAL: NCT04498715
Title: An Open-labelled Pilot Study to Evaluate Dynamic Hip Screw System (DHS) Augmented With a Biphasic Apatite Sulphate Combined With Systemic or Local Bisphosphonate for Trochanteric Femur Fracture
Brief Title: Trochanteric Femur Fracture Operated With Dynamic Hip Screw System (DHS) Augmented With a Biphasic Apatite Sulphate Combined With Systemic or Local Bisphosphonate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Lund University Hospital (Other)
Responsible Party: Principal Investigator, Sarunas Tarasevicius, Professor, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200723; Lithuanian (Other: Lithuanian University of Health Sciences)
Record Dates: First submitted 2020-07-27; First posted 2020-08-04 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Trochanteric Fracture of Femur
Keywords: Dynamic hip screw (DHS); Biphasic apatite sulphate ceramic; bisphosphonate-zoledronic acid
MeSH Terms: interventions — Fracture Fixation, Internal; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OSTEOSYNTHESIS+SYSTEMIC ZOLEDRONIC ACID (Active Comparator): After osteosynthesis, systemic Zoledronic acid 4mg (or any other bisphosphonate) will be given intravenously between day 7-14 post operation.
  Interventions: Procedure: OSTEOSYNTHESIS; Drug: Zoledronic Acid
- OSTEOSYNTHESIS+LOCAL CERAMENT BONE VOID FILLER (BVF)+SYSTEMIC ZOLEDRONIC ACID (Experimental): During osteosynthesis, cerament BVF will be used for the augmentation of the screw. Then systemic Zoledronic acid 4mg (or any other bisphosphonate) will be given intravenously between day 7-14 post operation.
  Interventions: Procedure: OSTEOSYNTHESIS; Drug: Zoledronic Acid; Device: CERAMENT BONE VOID FILLER (BVF)

INTERVENTIONS:
Procedure: OSTEOSYNTHESIS — Routine procedure for anesthesia and infection prophylaxis according to the clinics routines will be followed. The patient is supine with the fractured leg positioned in traction table. The biplanar x-ray device is moved and adjusted for proper simultaneous AP and lateral view. Hip region is washed and dressed in sterile draping's. Using standard proximal femur osteosynthesis technique 2.0 mm diameter Kirschner wire is placed in the middle zone of the femoral neck in AP and lateral view. The canal is opened using 6 mm drill bit and measured length of dynamic hip screw is placed in the femoral head and neck.
Drug: Zoledronic Acid — Zoledronic acid (ZA), is a bisphosphonate, and has been shown to reduce the risk of hip fracture by 41% in post-menopausal women. For systemic injection, 4 mg (as per clinical protocol) will be injected intravenously 1-2 weeks after surgery. For local delivery, 1 or 2 mg Zoledronic Acid will be added to 5 or 10 mg CERAMENT BVF during mixing and the mixture will be injected.
  Other Names: Zometa
Device: CERAMENT BONE VOID FILLER (BVF) — CERAMENT™|BONE VOID FILLER is a synthetic, injectable, osteoconductive bone void filler. CERAMENT™I is biphasic, consisting of 60% calcium sulfate and 40% hydroxyapatite mixed with the radio-opacity enhancing component CERAMENT™|C-TRU (iohexol 300 mg iodine/ml), which allows bone in-growth after curing. The high injectability of CERAMENT™ allows transcortical administration and ensures good intraosseous spread. In this trial, CERAMENT BVF paste will be injected by a sterilized metal needle (2-3 mm diameter and 15 cm length) through the hollow dynamic hip screw.
  Arms: OSTEOSYNTHESIS+LOCAL CERAMENT BONE VOID FILLER (BVF)+SYSTEMIC ZOLEDRONIC ACID

SUMMARY:
The purpose of this study is to study the process of bone regeneration around a metal device in the femoral neck canal using a synthetic bone substitute Cerament bone void filler (BVF) and bisphosphonate (Zometa) locally or systemically that affects bone metabolism. Furthermore, fracture healing and implant migration will be investigated.

DETAILED DESCRIPTION:
Osteoporosis associated fragility fractures in the elderly are a societal and financial burden in the western world and this burden has also started to affect developing nations. With the aging of the world's population, the age quake, hip fractures are expected to reach 2.6 million by the year 2025, and between 4.5 to 6.3 million by the year 2050. The mortality rate at 30 days after sustaining a hip fracture is up to 10%, and at one year 35% after the fracture. It is further known that almost half of the survivors are unable to reach their previous functional levels, partly related to the surgical treatment and fixation failure.

One fifth of all fragility fractures is in the hip with an almost equal ratio in in the cervical and trochanteric regions. Hip arthroplasty and internal fixation are the two most common treatment options for cervical and trochanteric femoral fractures. Healthier patients with long life expectancy have better functional recovery and lower mortality when internal fixation is used. However, dynamic hip screws (DHS) and intramedullary nails and screws are associated with high failure rates, particularly in unstable trochanteric fractures. Osteosynthesis cutout, with penetration of the cervical screw through the femoral head, preceded by a neck-shaft varus tilting, is the most common reason of failure, reported in up to 10% in trochanteric fractures, and in about 5% of neck fractures. In addition, reoperations have been reported to be as high as 30%, where treatment of dislocated femoral neck fracture with internal fixation fails and subsequently gets revised with total hip arthroplasty (THA). It is well established that salvage THA following hip fractures has significantly higher risk of complications compared to primary THA. The tip-apex distance has been defined as a strong predictor of screw cutout, while recent studies question its relevance. The bone quality, i.e. the degree of osteoporosis, on the other hand is associated with failures.[4] Despite the increase in clinical awareness; adoption of secondary prevention using bisphosphonates is still low, partly due to low patient adherence. Besides, even if included in a dual-energy X-ray absorptiometry surveillance program, there is a delayed response to bisphosphonate treatment, which has been deemed critical, during the first one and half years. Augmentation increasing mechanical strength of cancellous bone in osteoporotic hip fractures may lower the burden of revision, which may outweigh the related additional cost. Before the operation, deciding in whom to augment is a challenge A pilot study by Sirka et al. indicated that local delivery of a bisphosphonate, zoledronic acid (ZA), using the calcium sulphate/hydroxyapatite(CaS/HA) biomaterial enhanced bone formation in the femoral neck canal of severely osteoporotic rats. Moreover, recently, Raina et al. confirmed the findings also in a screw implant-integration model in rats. Whether these studies will show a similar potential in the clinical scenarios is a matter of speculation; however, they do provide novel methods for augmenting bone quality in osteoporosis as well as improving screw fixation. It is however important to mention that local delivery of ZA has a profound effect on cancellous bone regeneration in healthy as well as osteoporotic while the effect on cortical bone is minimal. A finite element modeling study by Kok et al. used computer simulations to predict the effect of CaS/HA augmentation in the form of injections into the human femoral heads/femoral neck canal and indicated enhanced mechanical properties by up to 25% which were dependent on volume and location of the injection. In a limited one-year follow up study, the use of an injectable ceramic applied in the trochanteric fracture bone void has been shown to lead to adequate fracture healing with minimal DHS screw migration Preliminary data from biomechanical studies in osteoporotic sawbones and donated human osteoporotic femoral heads indicates that using a biphasic apatite/sulphate material for reinforcing a fragile bone will result in an increase strength of the fixation of a fracture device inserted in the proximal femoral canal.(in house on file It is reasonable to argue that patients with high fracture and low mortality risks would benefit from an augmentation procedure far more than the ones with low fracture and high mortality risks. In a recent study, by combining the well-established fracture risk assessment tool (FRAX) and the Sernbo score to form a fracture and mortality risk evaluation (FAME) Index, one fifth of the patients could be identified as a cohort, with high risk of subsequent fracture but low risk of mortality. This group could theoretically benefit from cancellous bone augmentation during internal fixation of a fragility hip fracture. By utilizing a simple form, the FAME Index was successfully applied in the acute setting before the operation, during history taking by well-informed medical staff in less than 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients 65-90 years of age;
* Fame classification with low mortality and high fracture risk.
* Unilateral proximal hip fracture ((AO Foundation/Orthopaedic Trauma Association (AO/OTA): A1 and A2)) caused by low energy trauma (physical condition eligible for surgery with dynamic hip screw);
* Patient with a communicative ability to understand the procedure and participate in the study and the follow-up program.

Exclusion Criteria:

* Previous hip or pelvic fractures on the same side,
* Concurrent oral treatment with corticosteroids, and/or osteoporosis medication
* Irreversible coagulopathy or bleeding disorder. Note regarding reversible coagulopathies: Patients on coumadin or other anticoagulants may participate. Investigators should follow routine practices for perioperative discontinuation and re-initiation of anticoagulants;
* Concurrent dialysis or elevated creatinine
* Hypo or hyper calcaemia
* Active treatment due to malignancy including ongoing or completed radiotherapy involving the pelvis/hip area,
* Fractures involving acetabulum
* Active systemic infection or local skin infection at the incision site
* Known hyperthyroidism or thyroid adenoma,
* History of serious reaction to iodine based radio contrast agents

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change of bone density and remodeling around the head of dynamic screw | 1.5, 3, 6 months
  Bone density and remodelling around a dynamic hip screw will be investigated by CT scan using a program for alleviating metal artefacts. A 20% increase in bone density is expected to be significant and clinically relevant.

SECONDARY OUTCOMES:
Change of Harris Hip Score (HHS) in different group patients | 1.5, 3 and 6 months
  The HHS score has a maximum of 100 points (best possible outcome) covering pain (1 item, 0-44 points), function (7 items, 0-47 points), absence of deformity (1 item, 4 points), and range of motion (2 items, 5 points). The higher the HHS, the less dysfunction. A total score of <70 is considered a poor result; 70-80 is considered fair, 80-90 is good, and 90-100 is an excellent result.
Change of the Screw migration by X-ray | 1.5, 3 and 6 months
  Quantify dynamic hip screw (DHS®) migration on serial anteroposterior (AP) radiographs by accounting for femoral rotation and flexion.

CONTACTS AND LOCATIONS:
Overall Officials: Sarunas Tarasevicius, MD,PhD, Principal Investigator — Lithuanian University of Health Sciences
Locations (1):
- Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared after the study finished.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 5-10 years after study finished.
Access Criteria: Universities, hospitals and research institutions.

REFERENCES:
- [Result] Raina DB, Markeviciute V, Stravinskas M, Kok J, Jacobson I, Liu Y, Sezgin EA, Isaksson H, Zwingenberger S, Tagil M, Tarasevicius S, Lidgren L. A New Augmentation Method for Improved Screw Fixation in Fragile Bone. Front Bioeng Biotechnol. 2022 Mar 2;10:816250. doi: 10.3389/fbioe.2022.816250. eCollection 2022. PMID 35309986
- See also: Related Info — https://doi.org/10.3389/fbioe.2022.816250